CLINICAL TRIAL: NCT03373799
Title: Effectiveness of Video-Based Rehabilitation Program on Pain, Functionality and Quality of Life in the Treatment of Rotator Cuff Tears
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Ezgi Türkmen, Research Assistant, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IstanbulU30
Record Dates: First submitted 2017-11-25; First posted 2017-12-14 (Actual); Last update posted 2017-12-14 (Actual); Status verified 2017-12

CONDITIONS: Rotator Cuff Tear; Pain, Shoulder
Keywords: rotator cuff; physiotherapy; video-based rehabilitation; exercise
MeSH Terms: conditions — Rotator Cuff Injuries; Shoulder Pain; Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Video-Based Rehabilitation Group
  Interventions: Other: Video-Based Rehabilitation Program
- Group 2 (Active Comparator): Physiotherapist-Supervised Rehabilitation Group
  Interventions: Other: Physiotherapist-Supervised Rehabilitation Program

INTERVENTIONS:
Other: Video-Based Rehabilitation Program — In both groups, a program consisting of exercises used in conservative treatment of rotator cuff tears was performed. A video record was made by the physiotherapist to a patient where each exercise was described in detail and the patient correctly performed the exercises according to the verbal and visual commands of the physiotherapist. This video record watched by the patients who come to the clinic and patients were asked to do the exercises in the video. Patients did the exercises under control of the physiotherapist in the clinic.
  Arms: Group 1
Other: Physiotherapist-Supervised Rehabilitation Program — In both groups, a program consisting of exercises used in conservative treatment of rotator cuff tears was performed. Program was carried out by teaching the same exercises individually by the physiotherapist.
  Arms: Group 2

SUMMARY:
The aim of this study was to investigate the efficacy of the video-based rehabilitation program on pain, functionality and quality of life in the conservative treatment of partial tears of the rotator cuff whether it was as successful as the physiotherapist-supervised rehabilitation program.

DETAILED DESCRIPTION:
In our study a common exercise program, which can be used in conservative treatment of a partial rotator cuff tear, is applied with two different methods; a video-based rehabilitation program and physiotherapist-supervised rehabilitation program. Video-based rehabilitation program was developed to investigate whether this program is effective on pain, functionality and quality of life and as successful as a physiotherapist-supervised rehabilitation program.

ELIGIBILITY:
Inclusion Criteria:

* Forty years of age or older patients that had been diagnosed for a partial rotator cuff tear that was unrelated to trauma by a specialist orthopedist with MRI and physical examination and no other shoulder problems on the diagnosed shoulder were included into this study.

Exclusion Criteria:

* Patients that had been diagnosed for a full-thickness or massive rotator cuff tear, operated previously, had frozen shoulder or glenohumeral instability
* Younger than 40-year-old, and athletic patients with acute tear symptom were excluded from this study.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2016-05-30 (Actual); Primary Completion 2017-03-30 (Actual); Study Completion 2017-03-30 (Actual)

PRIMARY OUTCOMES:
Shoulder Range of Motion (ROM) | Shoulder range of motion evaluation was performed first time at baseline and second time after 6 weeks rehabilitation program. After treatment "change" was assessed.
  The shoulder flexion, abduction, internal and external rotation ROM were evaluated with goniometer while the patient was in supine position.

SECONDARY OUTCOMES:
Visual Analogue Scale (VAS) | Evaluation was performed before treatment and after 6 weeks rehabilitation program. Patients were asked to evaluate their pain status with a 10-point scale and high scores are positively correlated with pain.
  The levels of pain felt at rest / activity / night were measured using visual analogue scale (VAS).
ASES (The American Shoulder and Elbow Surgeons Standardized Shoulder Assessment) Form | Evaluation was performed before treatment and after 6 weeks rehabilitation program.
  ASES is an assessment form prepared by shoulder and elbow surgeons with objective and subjective sections. The total score is at least 0 and at most 100, and the high scores are positively correlated with the normal function.
Disabilities of the Arm, Shoulder and Hand (DASH) Questionnaire | Evaluation was performed before treatment and after 6 weeks rehabilitation program.
  DASH questionnaire inquires about the activities of a person in daily life, the degree of participation in recreational activities, the symptom and psychosocial state that affects their pain, emotional state and sleep quality. The total score is at least 0 and at most 100, and the high scores are positively correlated with the increased functional impairment.
Short Form 12 (SF-12) | Evaluation was performed before treatment and after 6 weeks rehabilitation program.
  SF-12 was used to assess physical and mental health-related quality of life. The total score is at least 0 and at most 100, and the high scores are positively correlated with high quality of life.
Global Rating of Change (GRC) Scale | Evaluation was performed after 6 weeks rehabilitation program.
  Global Rating of Change (GRC) scale was used to assess the overall satisfaction levels of the patients. Patients were asked to evaluate their post-treatment status with a 5-point likert scale and high scores are positively correlated with satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Ezgi Türkmen, Principal Investigator — Istanbul University
Locations (1):
- Istanbul University, Istanbul, Bakırkoy, Turkey (Türkiye)